CLINICAL TRIAL: NCT06014931
Title: Telehealth-enhanced Patient-oriented Recovery Trajectory After Intensive Care
Acronym: TelePORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Ohio State University (Other)
Responsible Party: Principal Investigator, Leanne M Boehm, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 190790-Phase 2; R01AG077644 (NIH)
Record Dates: First submitted 2023-08-01; First posted 2023-08-28 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Post-intensive Care Syndrome
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telemedicine ICU Recovery Clinic (Experimental): scheduled telemedicine study visits 3 weeks and 3 months after hospital discharge or return-to-home if discharged to another facility
  Interventions: Behavioral: Telemedicine ICU Recovery Clinic Visit
- Standard Recovery Conditions (i.e., Control) (No Intervention): Control group participants will proceed with follow-up as determined by the discharging hospital team and directed to use the provided PICS guide to connect with commonly used resources.

INTERVENTIONS:
Behavioral: Telemedicine ICU Recovery Clinic Visit — Multidisciplinary clinic visit that encompasses a medical examination, medication management, neuropsychological exam with focused psychotherapy, case management, and patient-centered consultation.
  Arms: Telemedicine ICU Recovery Clinic

SUMMARY:
Intact cognitive skills are necessary for independent living, going to work, and managing finances, and any loss of cognitive skills places a burden on society akin to what is seen with Alzheimer's Disease and Related Dementias. The TelePORT Study (Telehealth-Enhanced Patient-Oriented Recovery Trajectories after Intensive Care) is the first post-intensive care syndrome longitudinal long-term cognitive impairment intervention study. The societal effect from long-term cognitive impairment after critical illness is great as many of these patients are employable adults or functional retirees.

DETAILED DESCRIPTION:
Up to 80% of Intensive Care Unit (ICU) survivors experience cognitive, physical, mental, and socioeconomic impairments, known as Post-Intensive Care Syndrome (PICS), that can last months to years following critical illness and lead to significant reductions in quality of life. Among historical cohorts of acute respiratory distress syndrome and sepsis survivors, as many as 80% demonstrate PICS-related acquired dementia. Likewise, in a broad group of ICU survivors in all adult age groups, 33% to 50% have acquired dementia. ICU Recovery Clinics (ICU-RC) are a feasible and promising intervention to address multifactorial PICS impairments collaboratively, but in-person access is limited. There is an unmet need to study the efficacy of clinics with large cohorts that apply alternative delivery strategies to enhance availability and reach. Older adult (age >=45) ICU survivor is at a combined risk for long-term cognitive impairment (LTCI) among other PICS impairments, and the ideal population to first address this knowledge gap. The investigators hypothesize that a collaborative telemedicine-delivered interdisciplinary ICU-RC intervention effectively identifies and improves LTCI, physical and mental health dysfunction, social integration, and self-management behaviors vs. a control condition with follow-up chosen by the discharge team. Therefore, in a sample of older septic shock and acute respiratory failure survivors, the investigators aim to examine the efficacy of telemedicine ICU-RC services vs. control follow-up chosen by the discharge team in identifying PICS impairments and improving cognitive, physical, and mental health function; and social integration and self-management behaviors at 6 months after hospital discharge. This willl be achieved via a randomized controlled trial of 202 patients randomized 1:1 with age stratification to telemedicine ICU-RC or control (101 per group). Telemedicine recipients will receive a minimum of 2 ICU-RC visits within 3 months of hospital discharge or return to home if discharged to another institution, with additional follow-up determined by the severity of PICS impairment. Cognitive, mental health, and physical outcomes will be measured using the Long-term Core Outcome Measurement Set for ICU survivors in addition to the Social Network Index and Patient Activation Measure. Measures are timed to assess pre-hospital, 1-week post-discharge, and 6-month post-discharge functioning trajectories. This research will provide scientific justification for the continued development, implementation, and scaling of ICU recovery care programs. Ultimately, such knowledge can improve the quality of life for millions of ICU survivors and their family members.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥45)
* Admitted to a medical or surgical ICU
* Treated for ARF (with mechanical ventilation) and/or septic shock (with vasopressors)

Exclusion Criteria:

* hospice care at discharge or not expected to survive 6 months
* no access to a computer or electronic device (e.g., tablet, smart phone) with cellular or WiFi connection for a telemedicine clinic visit
* substance abuse or psych disorder that prevents independent living
* inability to speak English
* severe dementia preventing independent living prior to index hospitalization

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive function - MoCA | 6 months
  The Montreal Cognitive Assessment-Blind is a 13-item widely used research measure for cognitive function that assesses memory, attention, language, recall, orientation, and abstraction. Test scores range from 0 (worst) to 22 (best) with a score below 18 being abnormal. Individual tasks on the MoCA-Blind are relatively difficult, reflecting less of a ceiling effect than comparable tools. Among widely used global screening measures, the MoCA has been consistently found to be the most sensitive in identifying even mild expressions of cognitive impairment.
Cognitive function - PROMIS | 6 months
  The PROMIS Cognitive Function is an 8-item patient-reported outcome measure assessing patient-perceived changes in mental acuity, verbal/nonverbal memory, verbal fluency, and concentration. Raw scores are converted to a standardized T-score with a mean of 50. Higher T-scores indicates better cognitive function.

SECONDARY OUTCOMES:
Physical function - ADL | 6 months
  Katz's Activities of Daily Living (ADL) is a 6-item self-report of ability to perform ADLs (e.g., bathing, dressing) independently. Items are scored as 0 (dependent) or 1 (independence). Summary scores range from 0-6 with lower scores indicating greater dependence.
Physical function - IADL | 6 months
  Lawton's Instrumental Activities of Daily Living (IADL) is an 8-item self-report of independence in performing IADLs (e.g., meal preparation, finance management). Items are scored as 0 (dependent) or 1 (independence). Summary scores range from 0-8 with lower scores indicating greater dependence.
Physical function - quality of life | 6 months
  EuroQol-5D-5L is a 6-item self-report questionnaire of health status. Items are scored on 5 levels of severity ranging from 'no problems' to 'extreme problems' and higher scores indicating worse quality of life.
Mental health - PTSD | 6 months
  PTSD symptoms will be measured using the Impact of Events Scale-Revised (IES-R), a 22-item tool designed to measure the subjective distress caused by traumatic events. Subjects rate each item from 0 (not at all) to 4 (extremely) to indicate the degree to which they have been bothered by a particular symptom over the past week. Total score is obtained by calculating the mean of all items. Subscale scores can be calculated for avoidance, hyperarousal, and intrusion. Higher scores indicate more distress related to the specific event being evaluated.
Mental health - anxiety/depression | 6 months
  Depression and Anxiety will be measured using the Hospital Anxiety and Depression Scale (HADS), a 14-item self-report. Subjects rate each item from 0 (absence) to 3 (extreme) to indicate the degree to which they have experienced the symptom in the past 7 days. The total possible score ranges from 0-21 per subscale with more than 11 being abnormal.
Social integration | 6 months
  Berkman-Syme's Social Network Index measure of marital status, friends/family contact, church membership, and group membership. The index considers number and importance of social ties across categories using a summative measure (range: 0-4). For example, there is heavier weighting for intimate contacts (4x the weight of group membership) over church membership (2x the weight of group membership).
Self management | 6 months
  Patient Activation Measure, a 13-item survey quantifying how much someone is informed about and involved in their health care. The raw score is converted to an activation score (range: 0 [no activation] to 100 [high activation]). Domains assess importance of active role, confidence and knowledge to take action, taking action, and continuing healthy behaviors under stress.

OTHER OUTCOMES:
Post-Traumatic Growth | 6 months
  Post-Traumatic Growth Inventory, a 21-item scale with higher scores indicating greater post-traumatic growtth

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Boehm, PhD, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Sharing data generated by this project is an essential part of the proposed research. The investigators seek to make data available to the community of scientists interested in ICU recovery care, specifically related to older adults attending ICU-RCs. The TelePORT trial will yield longitudinal outcomes data from approximately 202 adults. The final data set will contain de-identified demographic information and patient outcome responses on PICS, social integration, self-management, and other exploratory outcomes. Data will be available for sharing after the publication date of the main results from the final dataset.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after study completion
Access Criteria: When approval is granted, data-sharing agreements that provide for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed will be instituted. Requests for data must be made in writing and must clearly state the intended use of the requested data and expected length of time for data analyses. This request must be sent directly to the study contact PI who will record all requests for NIH reporting and secure IRB involvement in the process.

REFERENCES:
- [Background] Boehm LM, Danesh V, Eaton TL, McPeake J, Pena MA, Bonnet KR, Stollings JL, Jones AC, Schlundt DG, Sevin CM. Multidisciplinary ICU Recovery Clinic Visits: A Qualitative Analysis of Patient-Provider Dialogues. Chest. 2023 Apr;163(4):843-854. doi: 10.1016/j.chest.2022.10.001. Epub 2022 Oct 13. PMID 36243061
- [Background] Boehm LM, Danesh V, LaNoue M, Trochez RJ, Jones AC, Kimpel CC, Sevin CM. Factors Influencing Engagement with in-Person Intensive Care Unit Recovery Clinic Services. J Intensive Care Med. 2023 Apr;38(4):375-381. doi: 10.1177/08850666221127154. Epub 2022 Sep 21. PMID 36128790
- See also: PI profile — https://nursing.vanderbilt.edu/people/bio/leanne-boehm
- See also: Vanderbilt ICU Recovery Center — https://www.icudelirium.org/the-icu-recovery-center-at-vanderbilt